CLINICAL TRIAL: NCT02755207
Title: Potential Diagnostic and Prognostic Value of microRNAs for the Patients of Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Bin He, M.D./Ph.D., Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-003
Record Dates: First submitted 2016-03-29; First posted 2016-04-28 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2019-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Suspected ACS group: Patients admitted to the hospital with the diagnosis of ACS
- Blank control group: Patients admitted to the hospital without the diagnosis of ACS

SUMMARY:
The purpose of this study is to evaluate the potential diagnostic and prognosis value of circulating microRNAs compared with cTnI for suspected ACS patients at the emergency department (ED) and intensive care unit (ICU).

DETAILED DESCRIPTION:
The present study is a single-center, prospective diagnostic study among patients presenting to the ED or ICU within 24 h of onset of chest pain suggestive of suspected ACS.

We propose to construct the biobank of ACS and evaluate the potential diagnostic value of circulating microRNAs compared with cTnI for suspected ACS patients. All the patients are to be followed up for 6 months. Final diagnosis was made by an expert panel cardiologist, based on all available clinical information including cTnI measurements, ECG, coronary angiography, cardiac exercise tests and information from hospital discharge letters.

The concentrations of microRNAs will be evaluated by quantitative reverse transcription PCR, using highly specific primers and hybridization probes.

ELIGIBILITY:
Inclusion Criteria:

Suspected ACS patients (STEMI, NSTEMI, and UA):

Age>18 years; Informed consent.

Exclusion Criteria:

Patients who will undergo immediate PCI; Pregnant and lactating women; Patients with mental disorders; Patients are using other experimental drugs; Refusal to provide informed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Suspected ACS patients (STEMI, NSTEMI, and UA)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic value of microRNAs in qPCR，in ACS | Day 7

SECONDARY OUTCOMES:
Evaluate the prognostic value of microRNAs in ACS | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided